CLINICAL TRIAL: NCT06253780
Title: Multidisciplinary Study to Verify Blood Pressure Documentation and Response to Titration of Intravenous Medications
Acronym: VERBATIM
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Principal Investigator, DaiWai Olson, Professor, University of Texas Southwestern Medical Center
Other Study IDs: 3034
Record Dates: First submitted 2024-01-30; First posted 2024-02-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure
Keywords: neurovascular illness; Neurocritical care; Blood pressure; Continuous data acquisition; Neurology; Neurosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Adult patients (age > 18 years old) admitted to the NSICU at UT Southwestern Medical Center with a neurological, neurosurgical, or neurovascular diagnosis are eligible receiving Intravenous vasoactive medication infusing at the time of consent.

SUMMARY:
This study is an observational, non-randomized, study that will examine the variability in blood pressure (BP) response to intravenous (IV) vasoactive medications when BP is continuously sampled versus real-world BP sampling. Continuous BP sampling will be obtained using the Component Neuromonitoring System (CNS-200; Natus Corp) to obtain continuous data acquisition (CDA). The investigators will explore BP change based on electronic medical record (EMR) vs CNS-200 data. This study will consent and observe 30 Neuroscience Intensive Care Unit subjects using pragmatic sampling. Each subject will be observed one-and-only-one time for a 12-hour period.

DETAILED DESCRIPTION:
In this study, the investigators seek to explore if patients who receive continuous IV vasoactive medication infusion have a difference in blood pressure (BP) response measured and reported continuously versus intermittently. Adult patients (age > 18 years old) admitted to the Neuroscience Intensive Care Unit at The University of Texas Southwestern Medical Center with a neurological, neurosurgical, or neurovascular diagnosis are eligible. Patients must be receiving Intravenous vasoactive medication infusing at the time of consent. Eligible patients must have an indwelling Arterial line as placed as part of standard of care. There are no restrictions on obtaining Non-invasive BP during data collection. Patients, or legally authorized representatives (LARs), must be able to consent themselves in English. Subjects will be excluded if they are: Under the age of 18, pregnant, or they are currently incarcerated. Because the study does not have the availability to develop foreign language consents, subjects (or LARs) who are unable to read and communicate in English will also be excluded. The primary null hypothesis is that continuously acquired data from the arterial line have a similar mean and standard deviation as documented values in the EMR. The first step in examining this hypothesis is a simple paired T-test. An F-test will be used to compare the standard deviations. Rejection of the null will indicate the need for additional models to compare the median, Interquartile range (IQR), minimum and maximum values. The area under the curve will be determined as a function of the time above or below the prescribed BP range and the time spent outside of that range.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Admitted to the NSICU at UT Southwestern Medical Center with a neurological, neurosurgical, or neurovascular diagnosis
* Patients must be receiving Intravenous vasoactive medication infusing at the time of consent
* Eligible patients must have an indwelling A-line as placed as part of standard of care
* Patients, or legally authorized representatives, must be able to consent themselves in English.

Exclusion Criteria:

* Under the age of 18
* Pregnant
* Incarcerated upon admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study personnel will identify NSICU patients who are receiving an IV vasoactive medication infusion and are scheduled to have an arterial line (A-line) placed, or already have an A-line placed. This information is found in the EMR. Following consent, the study team will assign each patient a subject identification number (SID) that will be used as an alternate to any protected health information (PHI). After consent has been given, the study team will coordinate a time to place the CNS-200 monitor in the room of the patient. In the NSICU, the SOC is to routinely test BP using a cuff and or A-line.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Reported blood pressure reliability | 12-hour monitoring session once per enrolled patient (baseline)
  This study is an observational, non-randomized, study that will examine the variability in blood pressure (BP) response to intravenous vasoactive medications when BP is continuously sampled versus real-world BP sampling. Continuous BP sampling will be obtained using the Component Neuromonitoring System (CNS-200; Natus Corp) to obtain Continuous data acquisition (CDA) data. The investigators will explore BP change based on Electronic Medical Record (EMR) vs CNS-200 (CDA) data.

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, PhD, RN, FNCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States